CLINICAL TRIAL: NCT02804178
Title: A Phase 2, Multicenter Study of ATR-101 for the Treatment of Congenital Adrenal Hyperplasia
Brief Title: A Study of ATR-101 for the Treatment of Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millendo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATR-101-201
Record Dates: First submitted 2016-06-01; First posted 2016-06-17 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: ATR-101; classic congenital adrenal hyperplasia; 21-hydroxylase deficiency; CAH
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Congenital adrenal hyperplasia due to 21 hydroxylase deficiency | interventions — N-(2,6-bis(1-methylethyl)phenyl)-N'-((1-(4-(dimethylamino)phenyl)cyclopentyl)methyl)urea hydrochloride

STUDY DESIGN:
Intervention Model Description: Single treatment arm with up to 5 planned dosing periods with escalating doses. Subjects were dosed with each dose level for 2 weeks, followed by 2 weeks of matching placebo (subjects blinded).
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATR-101 (Experimental): Ascending dose levels of ATR-101 beginning with 125 mg by mouth twice per day up to 1000 mg twice per day.
  Interventions: Drug: ATR-101

INTERVENTIONS:
Drug: ATR-101 — 125-1000 mg twice per week
  Other Names: Nevanimibe hydrochloride

SUMMARY:
This is a Phase 2 multicenter, single-blind, multiple dose study to evaluate the safety and efficacy of orally administered ATR-101 in subjects with classic congenital adrenal hyperplasia (CAH). Treatment duration will range from a minimum of approximately 2 months to 6 months per subject. A subject may receive a minimum of one dose level or up to a maximum of 5 dose levels, in sequentially increasing dose strengths. Each dose level will last 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Documented historical diagnosis of classic CAH due to 21-hydroxylase deficiency based on: Documented genetic mutation in the CYP21A2 enzyme consistent with a diagnosis of classic CAH, or historical documentation of elevated 17-hydroxyprogesterone
* Biochemical marker of disease status of 17-hydroxyprogesterone ≥ 4 times the upper limit of normal
* Chronic glucocorticoid replacement therapy for at least 6 consecutive months
* Stable glucocorticoid and mineralocorticoid regimen for at least 1 month

Exclusion Criteria:

* Non-classic CAH
* Other causes of adrenal insufficiency
* Surgery within the previous 3 months prior to screening or planned surgery during study participation
* History of active cancer requiring medical or surgical therapy within the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - The University of Oklahoma - Tulsa Schusterman Center, Tulsa, Oklahoma
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Maouche D, Merke DP, Vogiatzi MG, Chang AY, Turcu AF, Joyal EG, Lin VH, Weintraub L, Plaunt MR, Mohideen P, Auchus RJ. A Phase 2, Multicenter Study of Nevanimibe for the Treatment of Congenital Adrenal Hyperplasia. J Clin Endocrinol Metab. 2020 Aug 1;105(8):2771-8. doi: 10.1210/clinem/dgaa381. PMID 32589738

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATR-101
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | ATR-101
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
17-hydroxyprogesterone [Mean (Standard Deviation); unit: ng/dL] | 6591.0 (5371.80)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction of 17-hydroxyprogesterone to </= 2 Times the Upper Limit of Normal at Any Time Following 2 Weeks of Dosing With ATR-101
Description: 17-hydroxyprogesterone was measured predose in the morning at the beginning and end of each dose level.
Time Frame: Evaluated at baseline and day 15 of each dose level. Each subject will have up to 5 dose levels.
Measure: Count of Participants; unit: Participants
Arm/Group | ATR-101
Number analyzed (Participants) | 10
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the patient signed informed consent until 4 weeks after the last dose of active drug.
Arm/Group | ATR-101
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATR-101 (N=10)
Enteritis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATR-101 (N=10)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gingival recession (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (5)
Migraine (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritis generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
The small number of subjects analyzed as a result of the rarity of the disease (congenital adrenal hyperplasia).and the stage of the study (phase 2a)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-01-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT02804178/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT02804178/SAP_001.pdf